CLINICAL TRIAL: NCT00657007
Title: A Phase 1, Multi-Center, Double-Blind, Single and Double Dose-Escalation Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of LymphoStat-B™ (Monoclonal Anti-BLyS Antibody) in Subjects With Systemic Lupus Erythematosus
Brief Title: Phase 1 Study of Belimumab in Subjects With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: William Freimuth, MD, PhD/Vice President of Clinical Research, Immunology, Rheumatology and Infectious Diseases, Human Genome Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBSL01; Partial NIH grant M01 RR 00043
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): IV infusion over 2 hours
  Interventions: Biological: Placebo
- Belimumab 1 mg/kg (Experimental): 1 mg/kg IV infused over 2 hours
  Interventions: Biological: belimumab
- Belimumab 4 mg/kg (Experimental): 4 mg/kg IV infused over 2 hours
  Interventions: Biological: belimumab
- Beimumab 10 mg/kg (Experimental): 10 mg/kg IV infused over 2 hours
  Interventions: Biological: belimumab
- Belimumab 20 mg/kg (Experimental): 20 mg/kg IV infused over 2 hours
  Interventions: Biological: belimumab

INTERVENTIONS:
Biological: belimumab — 1. 1 mg/kg, IV (in the vein) once on Day 0, with a final evaluation at Day 84 (Cohort 1).
  2. 1 mg/kg, IV (in the vein) on Days 0 and 21, with a final evaluation at Day 105 (Cohort 5).
  Other Names: LymphoStat-B™; BENLYSTA
  Arms: Belimumab 1 mg/kg
Biological: belimumab — 1. 4 mg/kg, IV (in the vein) once on Day 0, with a final evaluation at Day 84 (Cohort 2).
  2. 4 mg/kg, IV (in the vein) on Days 0 and 21, with a final evaluation at Day 105 (Cohort 6).
  Other Names: LymphoStat-B™; BENLYSTA
  Arms: Belimumab 4 mg/kg
Biological: belimumab — 1. 10 mg/kg, IV (in the vein) once on Day 0, with a final evaluation at Day 84 (Cohort 3).
  2. 10 mg/kg, IV (in the vein) on Days 0 and 21, with a final evaluation at Day 105 (Cohort 7).
  Other Names: LymphoStat-B™; BENLYSTA
  Arms: Beimumab 10 mg/kg
Biological: belimumab — 1. 20 mg/kg, IV (in the vein) once on Day 0, with a final evaluation at Day 84 (Cohort 4).
  2. 20 mg/kg, IV (in the vein) on Days 0 and 21, with a final evaluation at Day 105 (Cohort 8).
  Other Names: LymphoStat-B™; BENLYSTA
  Arms: Belimumab 20 mg/kg
Biological: Placebo — 1. IV (in the vein) on Day 0 (Cohorts 1-4).
  2. IV (in the vein) on Days 0 and 21 (Cohorts 5-8).
  Arms: Placebo

SUMMARY:
The purpose of thie study is to evaluate the safety, tolerability, immunogenicity, pharmacokinetics and pharmacodynamics of belimumab (LymphoStat-B™)in subjects with SLE.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of SLE by ACR criteria
* Stable SLE disease activity
* On stable SLE treatment regimen
* History of measurable autoantibodies

Key Exclusion Criteria:

* Pregnant or nursing
* Received a non-FDA approved investigational agent within last 28 days
* Received cyclosporin, intravenous immunoglobulin (IVIG) or plasmapheresis within last 6 months
* Active lupus nephritis requiring hemodialysis, intravenous cyclophosphamide (Cytoxan™), or high-dose prednisone (> 100 mg/day) within last 6 months
* Active central nervous system (CNS) lupus requiring medical intervention within last 6 months
* History of renal transplant
* History of clinical evidence of an active significant acute or chronic diseases
* Have required management or hospitalization of any infection within last 4 weeks.
* History of hypogammaglobulinemia or IgA deficiency
* Have current drug or alcohol addiction
* History of or test positive at screening for HIV, Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-02; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, immunogenicity, pharmacokinetics and pharmacodynamics of belimumab in subjects with SLE. | Days 0-105

SECONDARY OUTCOMES:
To evaluate the effect of belimumab on clinical disease activity, total serum IgG (and IgM, IgA, IgE) and concentrations of peripheral mature B lymphocytes and plasmacytoid cells, and markers of SLE disease activity, including autoantibodies. | Days 0-105

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - University of California-Los Angeles, Los Angeles, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Northwestern University Medical School, Chicago, Illinois
  - Rush-Presbyterian-St Luke's Medical Center, Chicago, Illinois
  - The University of Chicago Hospital, Chicago, Illinois
  - The University of Michigan Health System, Ann Arbor, Michigan
  - SUNY Downstate Medical Center, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Hospital for Joint Diseases, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731
- [Derived] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605
- [Derived] Struemper H, Chen C, Cai W. Population pharmacokinetics of belimumab following intravenous administration in patients with systemic lupus erythematosus. J Clin Pharmacol. 2013 Jul;53(7):711-20. doi: 10.1002/jcph.104. Epub 2013 May 16. PMID 23681782
- [Derived] Furie R, Stohl W, Ginzler EM, Becker M, Mishra N, Chatham W, Merrill JT, Weinstein A, McCune WJ, Zhong J, Cai W, Freimuth W; Belimumab Study Group. Biologic activity and safety of belimumab, a neutralizing anti-B-lymphocyte stimulator (BLyS) monoclonal antibody: a phase I trial in patients with systemic lupus erythematosus. Arthritis Res Ther. 2008;10(5):R109. doi: 10.1186/ar2506. Epub 2008 Sep 11. PMID 18786258